CLINICAL TRIAL: NCT00344188
Title: Host Response to Infection and Treatment in Leishmania Infection of Humans
Brief Title: Diagnosis and Treatment of Leishmania Infections
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010238; 01-I-0238
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-04-09

CONDITIONS: Leishmaniasis; Skin Diseases, Parasitic; Euglenozoa Infections; Parasitic Diseases
Keywords: Cutaneous; Visceral; Leishmanial Infection; MucocutaneousLeishmaniasis; Natural History
MeSH Terms: conditions — Leishmaniasis; Skin Diseases, Parasitic; Euglenozoa Infections; Parasitic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: This population of patients are referred from their physicians both regionally and nationally.

SUMMARY:
This study will examine the natural history of Leishmanial infections and their treatments. It will provide an opportunity for NIAID staff to learn more about leishmaniasis and perhaps to improve diagnostic tests for these infections. Patients between 2 and 80 years of age with known or suspected leishmaniasis are eligible for this study.

Participants will have routine blood tests and a biopsy to confirm leishmanial infection. The biopsy procedure will be determined by the type of infection local cutaneous leishmaniasis (LCL), mucocutaneous leishmaniasis (MCL) or visceral leishmaniasis (VL). CL will be confirmed with a punch biopsy, in which a cookie-cutter type razor is used to remove a small circular piece of skin tissue. MCL will be confirmed using a thin flexible tube inserted into the nose. This tube is used to examine the nose and upper airway and to remove a tissue sample, if an affected area is seen. VL will be confirmed with either a bone marrow or liver biopsy or a splenic aspirate. For these procedures, a small tissue sample is withdrawn through a needle placed in the hipbone, liver or spleen, respectively. Some patients may also have a skin test for leishmaniasis similar to tuberculin skin testing.

Treatment and length of hospital stay are determined by the type of infection. CL may be treated with Pentostam, amphotericin, amphotericin B, itraconazole or ketoconazole; ML with amphotericin B, or encapsulated amphotericin; and VL with Pentostam or encapsulated amphotericin. Pentostam is infused daily for 18 to 28 doses, most as an outpatient. Blood is drawn 3 times a week for safety tests and an electrocardiogram is done 2 to 3 times a week to monitor heart rhythm. Amphotericin B is infused every day or every other day for about 30 doses, all on an inpatient basis. Patients undergo hydration (infusion of a large amount of fluid) just before and immediately after each infusion to protect the kidneys. Blood is drawn every other day and urine samples are collected occasionally for routine urinalysis. Encapsulated amphotericin is infused every other day, on an outpatient basis. Blood is generally drawn every other day to every 2 days and urinalyses are done periodically. Itraconazole and ketoconazole are taken orally for at least 1 to 3 months, with blood drawn every 2 to 3 weeks.

Patients may be asked to have photographs taken before, during and after treatment to document progress. They may also be asked to provide extra blood samples for research purposes, either through a vein in the arm or through apheresis, a method for collecting large numbers of cells. For apheresis, whole blood is collected through a needle in an arm vein and circulated through a machine that separates it into its components. The desired cells are then removed, and the rest of the blood is returned to the body, either through the same needle used to draw the blood or through a second needle in the other arm.

Patients with cutaneous leishmaniasis will have a follow-up clinic visit 2 weeks to 3 months after treatment is completed. If there are no complications, their participation will end at that time. Patients with mucocutaneous leishmaniasis and visceral leishmaniasis will be followed every 3 to 6 months indefinitely for routine evaluations and re-treatment if the infection recurs.

...

DETAILED DESCRIPTION:
Patients admitted on this protocol will have, or be suspected of having, a Leishmania infection. The major objectives of the protocol are to diagnose and classify the Leishmania infection and to provide species-based therapy to study the natural history of the treated infection and further understand host and species characteristics that lead to resistant or relapsing disease. As part of the standard evaluation of these patients, biopsies to obtain parasite and host tissue will be obtained. The host response before and after therapy will be assessed to address broader questions related to diagnosis, disease pathogenesis, and response to therapy. Careful observations of the patients clinical and immunologic responses to therapy will be made, as well as long-term follow-up of these changes. It is anticipated that the patients will receive optimal clinical care for their infections and that the specimens collected from them will prove to be valuable reagents for the laboratory studies of the host responses unique to leishmanial infections.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals aged 3 to 100 years.
* Diagnosis of leishmaniasis:

A: Biopsy proven

OR

B: Likely diagnosis of leishmaniasis based on :

Epidemiologic exposure, clinical manifestations, and time course

-Willingness to allow samples to be stored for future research.

EXCLUSION CRITERIA:

Any condition that, in the judgment of the investigator, may put the participant at undue risk or make them unsuitable for participation in the study.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This population of patients are referred from their physicians both regionally and nationally.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Estimated)
Dates: Start 2001-11-30 (Actual)

PRIMARY OUTCOMES:
Obtain phenotypic and clinical information to document refractory and relapsing clinical courses. | 1 year
  Obtain phenotypic and clinical information to document refractory and relapsing clinical courses.
Obtain organism genomic data at the initial time of NIH presentation and any further relapses | 1 year
  Obtain organism genomic data at the initial time of NIH presentation and any further relapses
Obtain a basic immune workup and host genetic information (WGS) | 1 year
  Obtain a basic immune workup and host genetic information (WGS)

SECONDARY OUTCOMES:
Assess the efficacy of varying treatment regimens in different species | 1 year
  Assess the efficacy of varying treatment regimens in different species
Assess the safety profile of varying treatment regimens | 1 year
  Assess the safety profile of varying treatment regimens

CONTACTS AND LOCATIONS:
Overall Officials: Elise M O'Connell, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-I-0238.html